CLINICAL TRIAL: NCT00507065
Title: A Phase III, Randomized, Multicenter, Double-blind, Parallel-Group, Placebo-Controlled Safety and Efficacy Study of ADDERALL XR With an Open Label Extension, in the Treatment of Adolescents Aged 13-17 With ADHD
Brief Title: Safety and Efficacy of ADDERALL XR in the Treatment of Adolescents Aged 13-17 With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLI381-314A
Record Dates: First submitted 2007-07-19; First posted 2007-07-25 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — SLI381

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Adderall XR (10 mg) (Experimental)
  Interventions: Drug: Mixed salts of a single-entity amphetamine (ADDERALL XR)
- Adderall XR (20 mg) (Experimental)
  Interventions: Drug: Mixed salts of a single-entity amphetamine (ADDERALL XR)
- Adderall XR (30 mg) (Experimental)
  Interventions: Drug: Mixed salts of a single-entity amphetamine (ADDERALL XR)
- Adderall XR (40 mg) (Experimental)
  Interventions: Drug: Mixed salts of a single-entity amphetamine (ADDERALL XR)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mixed salts of a single-entity amphetamine (ADDERALL XR)
  Arms: Adderall XR (10 mg); Adderall XR (20 mg); Adderall XR (30 mg); Adderall XR (40 mg)
Drug: Placebo
  Arms: placebo

SUMMARY:
Assess the safety and efficacy of ADDERALL XR compared to placebo in the treatment of adolescents (aged 13-17) with ADHD. Subjects were assigned to one of two cohorts based on weight (<= 75 kg or > 75 kg).

ELIGIBILITY:
Inclusion Criteria:

* Males/females 13-17 years of age meeting DSM-IV criteria for a primary diagnosis of ADHD

Exclusion Criteria:

* Controlled or uncontrolled comorbid psychiatric diagnosis (except ODD) with significant symptoms such as PTSD, psychosis, bipolar disease, severe OCD
* Known non-responder to stimulant medication
* Documented allergy or intolerance to ADDERALL, ADDERALL XR or amphetamines
* Conduct Disorder, hypertension, history of seizure
* Tic disorder or Tourette's disorder

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 329 (Actual)
Dates: Start 2003-05-28 (Actual); Primary Completion 2004-03-24 (Actual); Study Completion 2004-03-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline to final visit of the double-blind phase of the study in the ADHD-RS-IV score in the cohort weighing less than or equal to 75 kg. | approximately 4 weeks

SECONDARY OUTCOMES:
Change from baseline to final visit of double-blind phase of the study in ADHD-RS-IV score in the cohort weighing >75 kg and the CGI for ADHD in both cohorts. | Approximately 4 weeks
Adverse events, labs, physical exam, ECG | approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- New York University - Child Study Center, New York, New York, United States

REFERENCES:
- [Result] Spencer TJ, Wilens TE, Biederman J, Weisler RH, Read SC, Pratt R. Efficacy and safety of mixed amphetamine salts extended release (Adderall XR) in the management of attention-deficit/hyperactivity disorder in adolescent patients: a 4-week, randomized, double-blind, placebo-controlled, parallel-group study. Clin Ther. 2006 Feb;28(2):266-79. doi: 10.1016/j.clinthera.2006.02.011. PMID 16678648
- See also: FDA Recall information — http://www.fda.gov/opacom/7alerts.html